CLINICAL TRIAL: NCT00487812
Title: Prediction of Left Ventricular Remodelling in Patients Treated by Angioplasty in the Acute of Phase of a First Myocardial Infarction by Low-Dose Dobutamine Tc-99m-Mibi Gated SPECT
Brief Title: Low-Dose Dobutamine Tc-99m-Mibi Gated SPECT to Predict Left Ventricular Remodelling in Patients Reperfused in the Acute Phase of MI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Janusz LIPIECKI, CHU Clermont-Ferrand
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHU63-0017
Record Dates: First submitted 2007-06-18; First posted 2007-06-19 (Estimated); Last update posted 2008-10-07 (Estimated); Status verified 2008-10

CONDITIONS: Ischemic Heart Disease; Myocardial Infarction
Keywords: Acute myocardial infarction; left ventricular remodelling; SPECT imaging
MeSH Terms: conditions — Myocardial Ischemia; Myocardial Infarction

INTERVENTIONS:
Procedure: Low-dose dobutamine Tc-99-m-mibi gated SPECT imaging — All patients will be evaluated by ce-MRI during the initial hospital stay (5th - 6th day)

SUMMARY:
Left myocardial infarction (MI), has a negative impact of long term morbidity and mortality. Even in patients treated successfully by angioplasty in the acute phase of infarct, the remodelling is observed in approximately 30% of cases. It is important to predict the occurrence of this phenomenon in the early phase after MI for the selection of patients who could eventually benefit from new therapeutic approach as for example cell replacement therapy. It has been advocated that stem cells coronary injections should be performed between the 5th and 10th day after an acute event. We hypothesise that a low dose dobutamine gated Tc-99m-mibi SPECT performed on 5th-6th day after reperfused acute MI can predict left ventricular remodelling and serve as a method to screen patients who could benefit from cell replacement therapy.

DETAILED DESCRIPTION:
All patients will be evaluated by ce-MRI during the initial hospital stay (5th - 6th day) and at 6-month follow-up. Left ventricular remodelling will be defined as an end-diastolic volume increase of >20% between the two exams. A low dose dobutamine gated Tc-99m-mibi SPECT will be also performed on 5th-6th day. Differences in the infarct size and severity as well as the residual inotrope reserve in the infarct area are expected between groups with and without remodelling.

ELIGIBILITY:
Inclusion Criteria:

* Acute myocardial infarction,
* Successful coronary angioplasty in the acute phase,
* Absence of heart failure in the acute phase

Exclusion Criteria:

* acute heart failure in the acute phase
* severe ventricular arrhythmias
* contra indications for MRI imaging

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2004-12; Primary Completion 2006-08 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Development of left ventricular remodelling at 6-month follow-up | at 6-months follow-up

SECONDARY OUTCOMES:
Development of overt heart failure | development of overt heart failure

CONTACTS AND LOCATIONS:
Overall Officials: Lipiecki Janusz, Dr, Principal Investigator
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, Auvergne, France

REFERENCES:
- [Derived] Ernande L, Cachin F, Chabrot P, Durel N, Morand D, Boyer L, Maublant J, Lipiecki J. Rest and low-dose dobutamine Tc-99m-mibi gated-SPECT for early prediction of left ventricular remodeling after a first reperfused myocardial infarction. J Nucl Cardiol. 2009 Jul-Aug;16(4):597-604. doi: 10.1007/s12350-009-9098-5. Epub 2009 May 29. PMID 19479315